CLINICAL TRIAL: NCT02682407
Title: A Phase 2 Study to Evaluate the Safety and Effect on Proteinuria of OMS721 in Subjects With IgA Nephropathy, Lupus Nephritis, Membranous Nephropathy, or C3 Glomerulopathy Including Dense Deposit Disease
Brief Title: Safety Study of IgAN, LN, MN, & C3 Glomerulopathy Including Dense Deposit Disease Treated With OMS721
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS721-GNP-001
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: IgAN; Lupus Nephritis; MN; C3 Glomerulopathy
Keywords: IgAN; Lupus Nephritis; MN; C3 Glomerulopathy
MeSH Terms: conditions — Lupus Nephritis | interventions — narsoplimab

STUDY DESIGN:
Intervention Model Description: Cohort 2 and 3 subjects are randomized in a 1:1 fashion during the first 12 weeks of treatment. Cohort 1 and 4 are non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OMS721 (narsoplimab) (Experimental): Administration of OMS721 (narsoplimab)
  Interventions: Biological: OMS721 (narsoplimab)

INTERVENTIONS:
Biological: OMS721 (narsoplimab) — Biological: OMS721 (narsoplimab)
  Other Names: narsoplimab

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of OMS721 (narsoplimab) in subjects with Immunoglobulin A Nephropathy (IgAN), Lupus Nephritis (LN), Membranous Nephropathy (MN), and Complement Component 3 (C3) Glomerulopathy including Dense Deposit Disease. The study will also evaluate Pharmacokinetics (PK), Pharmacodynamics (PD), anti-drug antibody response (ADA), and neutralizing antibodies (NAb) of OMS721 when administered intravenously and when administered both intravenously and subcutaneously in subjects of Asian descent with IgA Nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening and competent to provide informed consent; For Cohort 4 only, participants are of Asian descent
* Have a diagnosis of one of the following:

  1. IgAN on kidney biopsy
  2. LN, MN and C3 Glomerulopathy including Dense Deposit Disease on kidney biopsy and 24-hour Urine Protein Excretion (UPE) > 1000 mg/24 hours (for Cohort 1 only)
  3. IgAN diagnosis is confirmed by biopsy within 8 years of screening for Asian descent (for Cohort 4 only)
* For Cohort 4 only: subjects with IgAN of Asian descent, documented history of 24-hour UPE > 1 g within 6 months prior to Screening or Urine Protein-Creatinine Ratio (uPCR) > 0.75 by spot urine at screening
* Screening Estimated Glomerular Filtration Rate (eGFR) >= 30 mL/min/1.73 m^2
* Are on physician-directed, stable, optimized treatment with angiotensin converting enzyme inhibitors (ACEI) and/or angiotensin receptor blockers (ARB) and have a systolic blood pressure of < 150 mmHg and a diastolic blood pressure of < 90 mmHg at rest

Exclusion Criteria:

* Have a hemoglobin less than 9.0 g/dL
* Have a platelet count =less than 100,000/mm^3
* Have an absolute neutrophil count <500 cells/mm^3
* Have an Alanine aminotransferase (ALT) or Aspartate Aminotransferase (AST) greater than 5.0 x the upper limit of normal (ULN)
* Have systemic manifestations of Henoch-Schonlein purpura within 2 years prior to Screening
* Have used: belimumab, eculizumab, or rituximab within 6 months prior to Screening
* Have a history of renal transplant
* History of human immunodeficiency virus (HIV), evidence of immune suppression, active hepatitis C virus (HCV) infection (subjects with positive anti-HCV antibody
* Have a malignancy except for adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or other cancer from which the patient has been disease-free for 5 years or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1-3: Proportion of IgAN, LN, MN, C3 Glomerulopathy subjects with treatment related adverse events (AE). | up to 104 weeks
Cohort 4: Proportion of IgAN patients of Asian descent with treatment related AEs. | 38 weeks
Cohort 4: Change from baseline in serum and urine complement component levels. | 38 weeks

SECONDARY OUTCOMES:
Cohort 1-3: Change from baseline in serum narsoplimab concentrations. | up to 104 weeks
Cohort 4: Change from baseline in serum narsoplimab concentrations. | 38 weeks
Cohort1-3: Change from baseline in proteinuria. | up to 104 weeks
Cohort1-3: Change from baseline in urine albumin/creatinine ratio. | up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Omeros Investigational Site, Denver, Colorado
  - Omeros Investigational Site, Augusta, Georgia
  - Omeros Investigational Site, Lawrenceville, Georgia
  - Omeros Investigational Site, Evergreen Park, Illinois
  - Omeros Investigational Site, Voorhees Township, New Jersey
  - Omeros Investigational Site, Flushing, New York
  - Omeros Investigational Site, San Antonio, Texas
  - Omeros Investigational Site, Milwaukee, Wisconsin
- Hong Kong (4):
  - Omeros Investigational Site, Chai Wan
  - Omeros Investigational Site, Hong Kong
  - Omeros Investigational Site, Kowloon
  - Omeros Investigational Site, Shatin